CLINICAL TRIAL: NCT03786224
Title: Pilot Trial on the Efficacy of Contingency Management for Six Months of Cannabis Abstinence Among Adolescents
Brief Title: Pilot Trial of Contingency Management for Long-Term Cannabis Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Randi Melissa Schuster, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018P001848
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: Cannabis Use; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abstinent (Experimental)
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Six months of cannabis abstinence will be incentivized using a standard contingency management approach involving an escalating schedule of payment for abstinence and attendance.

SUMMARY:
This study is a critically important first-of-its-kind investigation of the potential research utility of using contingency management to examine long-term changes in cannabis use with six months of abstinence. These pilot data will inform a later trial which will focus on testing the longitudinal relationships between adolescent cognition and cannabis use, questions of high and growing public health significance given adolescents' increased access to cannabis with legalization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents actively enrolled in a middle or high school in the Boston area who are between the ages of 13 and 19 (inclusive);
* Average use of cannabis at least 3 times per week during the 3 months prior to study enrollment;
* Cannabis use reported within 7 days of study enrollment;
* No immediate plan to discontinue cannabis use;
* Have a parent or legal guardian who is competent and willing to provide written informed consent for the active study phase (if under the age of 18);
* Competent and willing to provide written informed assent for the active study phase (if under the age of 18);
* Competent and willing to provide written informed consent (if age 18 or older);
* Able to communicate in English language;
* Have a parent/guardian who can communicate in English language;
* Able to commit to 27 study visits in approximately 6 months;
* Able to safely participate in the protocol and appropriate for outpatient level of care, in the opinion of the investigator.

Exclusion Criteria:

- Any severe developmental delays (including, but not limited to, Autism Spectrum Disorder, Intellectual Disability, and Down Syndrome).

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi M Schuster, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abstinent
Started | 6
Completed | 0
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Abstinent
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6
Urine THCCOOH [Mean (Standard Deviation); unit: ng/mL] | 281.9 (262.6)

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence Via Progressive Declines in Urine THCCOOH
Description: Cannabis abstinence will be indexed by progressively decreasing quantitative levels (ng/mL) of 11-nor-delta-9-THC-9-carboxylic acid (THCCOOH), the primary cannabis metabolite, in urine. Residual cannabinoid excretion will be differentiated from new cannabis exposure using a statistical model developed by Schwilke and colleagues (2011). This model was empirically derived from urine CN-THCCOOH concentration ratios of consecutively collected specimen pairs (current specimen/prior specimen). This model takes into account the time between collection of specimens, which enhances the accuracy of prediction of new cannabis use. This formula yields an expected CN-THCCOOH ratio associated with specimen pairs during abstinence, and observed ratios that exceed this expected value are interpreted as new cannabis use.
Time Frame: Six months
Population: 6 subjects enrolled in this pilot study and were included in the analysis. However, no participants completed data collection at the 6-month time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abstinent
Number analyzed (Participants) | 6
ng/mL | NA (NA) — No participants completed data collection at the 6-month time point.

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 6 months.
Description: Adverse events were collected at all study visits for all enrolled participants.
Arm/Group | Abstinent
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abstinent (N=6)
Loss of Appetitie (Metabolism and nutrition disorders) | 2 (8)
Skin Wound (Injury, poisoning and procedural complications) | 1 (2)
Indigestion (Gastrointestinal disorders) | 2 (2)
Common Cold (Infections and infestations) | 3 (5)
Worsening Depression (Psychiatric disorders) | 1 (1)
Worsening Suicidal Ideation (Psychiatric disorders) | 1 (1)
Increased Stress (Social circumstances) | 2 (10)
Difficulty Sleeping (General disorders) | 3 (15)
Soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Irritability (Psychiatric disorders) | 1 (4)
Hot flashes (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03786224/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03786224/ICF_001.pdf